CLINICAL TRIAL: NCT05365789
Title: A Trial to Evaluate Efficacy and Safety of a Nasal Spray Combined With Standard of Care for Nasal Congestion in Infants and Toddlers With Common Cold in Comparison to Standard of Care Alone
Brief Title: A Nasal Spray for Relief of Nasal Congestion in Infants and Toddlers With Common Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST-21-U58
Record Dates: First submitted 2022-01-27; First posted 2022-05-09 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Nasal Congestion
Keywords: Pediatric
MeSH Terms: conditions — Nasal Obstruction | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Open label, randomized, parallel group. Study product and standard of care versus standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Device and Standard of Care (Active Comparator): 1 to 2 sprays per nostril of Sterimar Blocked Nose Baby for a minimum of 2 times (morning and evening) and, as needed, up to a maximum of 6 times per day (i.e. maximum 12 sprays per nostril each day) until nasal symptoms are resolved, up to a maximum of 10 days.
  Standard of care consists of hydration, rest at home and antipyretic paracetamol as necessary.
  Interventions: Device: Blocked Nose Baby nasal spray; Other: Standard of care
- Standard of Care (Other): Standard of care consists of hydration, rest at home and antipyretic medication paracetamol as necessary.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Blocked Nose Baby nasal spray — One or two nasal sprays will be administered to each nostril for a minimum of 2 times per day up to a maximum of 6 times per day for a maximum of 10 days.
  Arms: Study Device and Standard of Care
Other: Standard of care — Standard of care consists of hydration, rest at home and antipyretic paracetamol as necessary.

SUMMARY:
The study will evaluate the safety and efficacy of the study medical device plus standard of care versus standard of care in subjects between 3 and 48 months (inclusive) presenting symptoms of a common cold.

DETAILED DESCRIPTION:
The purpose of the present study is to test the efficacy, safety and tolerability of a product in relieving the symptoms of the common cold in children. This nasal spray is specifically studied for small children, classified as medical devices and is already on the market. Sterimar Blocked Nose Baby (CDEU048-28) nasal spray is a medical device and is a 100 ml bag-on-valve spray. The spray contains hypertonic solution based on 100% natural sea water rich of marine trace elements with added manganese and copper.

220 subjects will be included in this open label, randomized, parallel group, study product and standard of care versus standard of care study.

Study product will be used as 1 to 2 sprays per nostril (each "dose" is 1 or 2 sprays per nostril, the second spray only if needed), for a minimum of 2 times (morning and evening) and, as needed, up to a maximum of 6 times per day (i.e., maximum 12 sprays per nostril each day). The 10 day study consists of 4 visits- Day 0 onsite, Days 3 and 6 telephone contact, and Day 10 onsite.

There will be 3 strata according to age: (3-12 months), (13-24 months) and (25-48 months). Every effort will be made to ensure at least 20% of subjects in each of the study groups are 3-12 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female infants and toddlers.
2. Aged 3 - 48 months (inclusive) at enrolment (Day 0).
3. Parent/legal guardian answering "yes" to the question "Do you feel that your child has a cold?" at enrolment.
4. Subjects with symptoms started not later than 48 hours prior to enrolment (Day 0).
5. Subjects with nasal congestion (blocked / stuffy nose) rated as at least score of 2 (moderately bothersome) on a 0 to 3-point scale, based on morning evaluation (within an hour of child awakening).
6. Subjects showing at least one of the following additional signs of cold symptoms: runny nose, nasal crust (dry mucus), thick mucus, sneezing and cough.
7. Parent/legal guardian of the subject has given freely and expressly her/his informed consent.
8. Parent/legal guardian is cooperative and aware of the necessity and duration of the controls so that perfect adhesion to the protocol established by the clinical trial center could be expected.

Exclusion Criteria:

1. Subjects presenting an oral temperature greater than 38°C at enrolment (Day 0).
2. Subjects presenting any secondary infection (such as bronchitis, otitis, tracheitis, pneumonia, etc.) at enrolment (Day 0).
3. Subjects with positive results on a streptococcal antigen screening test (rapid antigen detection test or RADT) at inclusion.
4. Subjects with a history of allergic rhinitis
5. Subjects presenting any congenital or chronic disease that in the opinion of the Investigator would adversely affect the results of the study (e.g. asthma, pneumonia, laryngotracheobronchitis, sinusitis, etc).
6. Subjects presenting any kind of immunodeficiency.
7. Subjects presenting any hypersensitivity or allergy or intolerance to any component of the study products or of the rescue medication (paracetamol)
8. Subjects with a positive medical history to any significant illness within the 2 weeks prior to the enrolment (Day 0).
9. Subjects presenting any active systemic infection or medical condition that may require treatment or therapeutic intervention during the study.
10. Subjects currently participating or having participated in another clinical trial during the last 30 days prior to enrolment (Day 0).
11. Subjects using saline nose drops or nasal sprays or pumps other than the study products, antibiotics, antivirals, intranasal medicines, decongestants, antihistamines, echinacea, combination cold formulas, supplements containing ≥ 10 mg zinc that would influence symptoms scores at enrolment (Day 0) within 12 hours prior the day of screening
12. Subject who was abroad in a country with a higher incidence rate of Covid-19 than Poland, within 14 days before the beginning of the study.
13. Subject who have had contact with any person infected with COVID-19 within 10 days before the beginning of the study.
14. Subject who are currently home quarantined, as recommended by the Sanitary Inspection.

Ages: 3 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change of nasal congestion | Through study completion, an average of 10 days.
  Assess reduction of nasal congestion, evaluated by means of a specific questionnaire ("Cold Symptom Severity Questionnaire") on a 0 to 3-point scale, with higher score indicating a worse outcome, with 0 =not at all, 1=mild, 2=moderate and 3=severe to be completed at Day 0 (baseline) and daily from the beginning to the end of the study; comparisons between groups.

SECONDARY OUTCOMES:
Change of other cold symptoms | Through study completion, an average of 10 days.
  Assess change of other cold symptoms, evaluated by means of a specific questionnaire ("Cold Symptom Severity Questionnaire"),on a 0 to 3-point scale, with higher score indicating a worse outcome, with 0=not at all, 1=mild, 2=moderate and 3=severe, to be completed at Day 0 (baseline) and daily from the beginning to the end of the study; comparisons between groups.
  Other cold symptoms: Stuffy nose, Nasal crust, Runny nose, Thick mucus, Sneezing, Cough
Occurrence of secondary infections | Through study completion, an average of 10 days.
  Assessment of occurrence of secondary infections (number) daily, from the beginning to the end of the study; comparison between groups. Secondary infections will be confirmed by the Investigator.

OTHER OUTCOMES:
Onset of relief | assessed at 5, 15, and 30 minutes post first application of device every morning from Day 0 to 3
  Assessment of onset of relief (immediate relief) after the entire product application is completed (1 or 2 sprays) at Day 0 (baseline) and daily from Day 1 to Day 3 of the study; within investigational device group.
  the study.
Concomitant medications | Through study completion, an average of 10 days.
  Assessment of use of concomitant medications (frequency, excluding paracetamol) will be done from the beginning to the end of the study; comparisons between groups.
Frequency of paracetamol administration. | Through study completion, an average of 10 days.
  Assessment of use of paracetamol (frequency) will be done from the beginning to the end of the study; comparisons between groups.
Quality of sleep. | Through study completion, an average of 10 days.
  Assessment of quality of sleep will be evaluated by means of a questionnaire ("Quality of Sleep Questionnaire"), on a 0 to 3-point scale, with higher score indicating a worse outcome, with 0=not at all, 1=slightly, 2=moderately and 3=severely, to be completed from Day 0 (baseline) and daily from the beginning to the end of the study; comparisons between groups.
Global assessment on common cold status. | Through study completion, an average of 10 days.
  Global assessment on common cold status will be evaluated by means of the "Global Assessment on Common Cold Status Questionnaire", on a 0 to 3-point scale, with higher score indicating a better outcome, with 0=no relief at all, 1=slight relief, 2=moderate relief and 3=complete relief, to be completed from the beginning to the end of the study; comparisons between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rynkiewicz, MD, Principal Investigator — Private Practice
Locations (1):
- PRIVATE PRACTICE ul. Osiedle Sierakowskich 5, Sztum, Poland

IPD SHARING:
Plan to Share IPD: Undecided